CLINICAL TRIAL: NCT03477383
Title: A New Biomarker for the Non-invasive Diagnosis of Rejection After Heart Transplantation
Acronym: BIODRAFT
Status: Completed | Type: Observational
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Lund University Hospital (Other); Karolinska University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ver 1.0; 014-16 (Other: Regional ethical review board in Gothenburg)
Record Dates: First submitted 2018-03-15; First posted 2018-03-26 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2021-10

CONDITIONS: Heart Transplant Rejection
Keywords: diagnosis; economics; cell-free DNA; digital droplet PCR; heart failure
MeSH Terms: conditions — Disease; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood plasma (10ml)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adult patients: Adult patients (18 years or older) undergoing heart transplantation
  Interventions: Diagnostic Test: donor-derived cell-free DNA (dd-cfDNA)
- Pediatric patients: Pediatric patients (0-17 years) undergoing heart transplantation
  Interventions: Diagnostic Test: donor-derived cell-free DNA (dd-cfDNA)

INTERVENTIONS:
Diagnostic Test: donor-derived cell-free DNA (dd-cfDNA) — Measurement of dd-cfDNA and comparison against grade of rejection as measured by endomyocardial biopsy, taken simultaneously

SUMMARY:
This study is a prospective, observational multi-center cohort study. The study will consist of patients undergoing heart transplantation. The main purpose is to test a new biomarker for rejection against the gold-standard, the endomyocardial biopsy (EMB). 80 patients will be included, both children and adults.

DETAILED DESCRIPTION:
The primary objective is a comparison of an the established, invasive diagnostic test, the endomyocardial biopsy (EMB) against a new, non-invasive test. The new test is the measurement of donor-derived cell-free DNA (dd-cfDNA) circulating in the blood stream of the recipient, quantified by droplet digital PCR (polymerase-chain reaction) after targeted multiplex preamplification. Sensitivity is calculated with EMB as the gold standard. The patients will be followed during one year post-transplantation with simultaneous blood samples and EMB. The patients will further be followed clinically for 5 years. A suitable cut-off for the ratio of dd-cfDNA will be calculated using receiver operating characteristic (ROC) analysis.

Secondary objectives are description of patient outcomes with respect to organ function, quality of life and adverse events.

Secondary objectives are the calculation of the costs related to the transplantation process as well as to the follow-up with EMB. A simulation will be done with respect to possible savings achieved if the new biomarker could be implemented.

The study consists of two cohorts: all adult recipients of heart transplantation at Sahlgrenska University Hospital (one of two center conducting heart transplantation in Sweden): regional study. The other cohort consists of all children undergoing heart transplantation in Sweden:national study. Patients will undergo transplantation at Sahlgrenska University Hospital in Gothenburg as well as at Skåne University Hospital in Lund. Follow-up with blood samples and EMB of these patients will be in Gothenburg, Lund and at Karolinska University Hospital in Stockholm.

ELIGIBILITY:
Inclusion Criteria:

1. Patient on waiting list for heart transplantation
2. Signed informed consent

Exclusion Criteria:

1. Follow-up outside Sweden

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients on waiting list for heart transplantion at the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Comparison of donor-derived cell-free DNA and endomyocardial biopsy with respect to rejection | 3 years
  Measurement of both fraction of donor-derived cell-free DNA of all cell-free DNA (derived from recipient and donor) as well as the absolute number of copies per ml plasma derived from the donor. Comparison is made with simultaneously obtained endomyocardial biopsies that are graded with respect to rejection, according to the official guidelines provided by the International Society of Heart and Lung Transplantation.

SECONDARY OUTCOMES:
Cost analysis 1 | 5 years
  Costs of heart transplantation during the first year post-transplantation
Rejection | 5 years
  Cumulative incidence of rejection (according to the biopsy grading system provided by the International Society of Heart and Lung Transplantation)
Graft-vasculopathy | 5 years
  Cumulative incidence of graft-vasculopathy
Overweight | 5 years
  Prevalence of overweight (BMI >25) and obesity (BMI>30)
Quality of life | 5 years
  Health-related quality of life as measured by EQ5D
Survival | 5 years
  Survival
Re-transplantation | 5 years
  Proportion of patients who have undergone re-transplantation
GFR (glomerular filtration rate) | 1 year
  Renal function evaluated by calculated and measured GFR (Iohexol or Cr-Clearance)
GFR (glomerular filtration rate) | 3 years
  Renal function evaluated by calculated and measured GFR (Iohexol or Cr-Clearance)
GFR (glomerular filtration rate) | 5 years
  Renal function evaluated by calculated and measured GFR (Iohexol or Cr-Clearance)
Infections | 5 years
  Cumulative incidence of infections requiring hospital admission
Circulatory support to transplantation | 5 years
  Proportion of patients undergoing heart transplantation from a ventricular assist device or extra-corporeal membrane oxygenation (ECMO) or from mechanical ventilation.
Immunization status | 5 years
  Impact of pre-transplantation immunization status on primary and secondary outcomes
Malignancy | 3 years
  Cumulative incidence of malignancy (post-transplantation lymphoproliferative disorder PTLD and others)
Malignancy | 5 years
  Cumulative incidence of malignancy (PTLD and others)
Prior cardiac surgery | 5 years
  Impact of prior cardiac surgery on other outcomes
Neonatal cardiac surgery | 5 years
  Impact of neonatal (first 4 weeks of life) cardiac surgery on other outcomes
Donor cardiac arrest | 5 years
  Correlation between circulatory arrest in the donor and cardiac function
Donor cardiopulmonary resuscitation (CPR) impact | 3 years
  Impact of CPR of the donor on the incidence of assumed early rejection
Initial immunosuppression | 5 years
  Correlation between initial immunosuppression and the incidence of rejection
Initial immunosuppression and malignancy | 5 years
  Correlation between type of initial immunosuppression and incidence of malignancy
Immunosuppression and adverse effects | 5 years
  Correlation of time points with over- or under-immunosuppression (as measured by blood levels of immunosuppressive drugs and comparison with desired levels) and the incidence of severe infection, renal function decline and malignancy
Immunosuppression and rejection | 5 years
  Correlation of time points with over- or under-immunosuppression (as measured by blood levels of immunosuppressive drugs and comparison with desired levels) with rejection events
Ischemia time | 5 years
  Correlation between ischemic graft time and cardiac function as measured by echocardiography
Blood products and adverse events | 5 years
  Correlation between the number of blood products (red blood cells, thrombocytes, plasma) given after transplantation and the incidence of adverse effects
Survival | 3 years
  Survival

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sunnegårdh, MD, PhD, Principal Investigator — Pediatric Heart Center, The Queen Silvia Children's Hospital, Sahlgrenska University Hospital
Locations (4):
- Sweden (4):
  - Transplantation Center, Sahlgrenska University Hospital, Gothenburg
  - Pediatric Heart Center, The Queen Silvia Children's Hospital, Sahlgrenska University Hospital, Gothenburg
  - Pediatric Heart Center, Skåne University Hospital, Lund
  - Pediatric Heart Center, Karolinska University Hospital, Stockholm

IPD SHARING:
Plan to Share IPD: Undecided
Not decided yet.

REFERENCES:
- [Derived] Bohmer J, Wasslavik C, Andersson D, Stahlberg A, Jonsson M, Wahlander H, Karason K, Sunnegardh J, Nilsson S, Asp J, Dellgren G, Ricksten A. Absolute Quantification of Donor-Derived Cell-Free DNA in Pediatric and Adult Patients After Heart Transplantation: A Prospective Study. Transpl Int. 2023 Oct 30;36:11260. doi: 10.3389/ti.2023.11260. eCollection 2023. PMID 37965628